CLINICAL TRIAL: NCT02122835
Title: Vascular and Metabolic Responses to Exercise Training in Heart Failure With or Without Type 2 Diabetes
Brief Title: Exercise, Heart Failure, and Type 2 Diabetes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding/patient availability
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00032063
Record Dates: First submitted 2014-04-18; First posted 2014-04-25 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2015-05

CONDITIONS: Heart Failure; Type 2 Diabetes
Keywords: exercise; aerobic exercise
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus, Type 2; Motor Activity

ARMS (2):
- heart failure (Other): aerobic exercise training
  Interventions: Behavioral: aerobic exercise training
- heart failure plus type 2 diabetes (Other): aerobic exercise training
  Interventions: Behavioral: aerobic exercise training

INTERVENTIONS:
Behavioral: aerobic exercise training — 12 weeks of supervised aerobic exercise training

SUMMARY:
The purpose of this study is to understand the differences in how patients with heart failure respond to exercise training compared to patients with heart failure and type 2 diabetes.

DETAILED DESCRIPTION:
The investigators will measure exercise capacity in patients with heart failure or heart failure plus type 2 diabetes prior to and following a 12-week exercise training program (5d/wk, 30 min/d, 60-75% VO2max) to determine whether improvements in exercise capacity in response to exercise training are mitigated in patients with combined heart failure plus type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* ≥50 yr of age
* New York Heart Association class II-III CHF and ejection fraction ≤35%
* receiving optimal medical therapy
* sedentary (≤ 30 min/wk structured physical activity).
* Half of volunteers (n=30) will have a diagnosis of type 2 diabetes (CHF+T2D).

Exclusion Criteria:

* smoking
* changes in medication ≤6 wk prior to enrollment
* major cardiovascular event or procedure ≤6 wk prior to enrollment
* foot ulcers
* advanced neuropathy
* co-morbidities or other limitations that may interfere with or prevent volunteers from safely completing the exercise training
* fixed rate pacemaker
* type 1 diabetes mellitus

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
exercise capacity | baseline, 12 weeks
  measured as peak oxygen consumption as well as treadmill time to exhaustion, also known as cardiopulmonary fitness

SECONDARY OUTCOMES:
flow-mediated dilation | baseline, 12 weeks
  brachial artery flow-mediated dilation
nitrite flux during exercise | baseline, 12 weeks
  changes in plasma nitrite during exercise

CONTACTS AND LOCATIONS:
Overall Officials: William Kraus, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States